CLINICAL TRIAL: NCT04708015
Title: A Retrospective Observational Clinical Study on the Use of Continuous Glucose Monitoring for Glycemic Control in Adult and Pediatric Patients With Glycogen Storage Disease Type Ia (GSDIa)
Brief Title: Retrospective Study of Glucose Monitoring for Glycemic Control in Patients With GSDIa
Status: Completed | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DTX401-CL001
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Glycogen Storage Disease Type IA
Keywords: Dexcom G6 iCGM; glucose metabolism disorder; CGM; Continuous Glucose Monitoring
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease; Glucose Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — A retrospective chart review of medical records

SUMMARY:
The primary objective of this study is to assess the percentage of time patients were in normal glucose control.

DETAILED DESCRIPTION:
Retrospective Dexcom G6 iCGM data stored in the Clarity cloud from eligible patients will be accessed and downloaded, stripped of patient-identifying information and provided to the contract research organization (CRO) to review prior to sending to the Sponsor for analysis of glycemic control. The CRO will ensure data shared with the Sponsor is de-identified and transferred over a secure file transfer platform. Further, Remote Site Specialists (RSSs) from the CRO will work with the healthcare providers (HCPs) from participating sites to obtain additional patient data including medical history, prescribed diet, cornstarch/Glycosade use and demographic data directly, if available, from the medical charts and will enter this information into an electronic data capture (EDC) system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GSDIa confirmed by either liver biopsy or molecular testing.
* Currently using the Dexcom G6 iCGM for glycemic control and with approximately one (1) month of CGM data available on the Dexcom Clarity cloud and have authorized sharing of data with thereferral center through the Dexcom Clarity app.

Exclusion Criteria:

* Presence or history of any disease, condition or chronic medication that, in the Investigator's opinion, would significantly affect interpretation of study results.
* Use of any investigational product or investigational medical device within 30 calendar days preceding screening or before completion of all scheduled study assessments during study enrollment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients eight years of age and older with GSDIa, who have used the Dexcom G6 iCGM for glycemic control, and with at least one month of CGM data available on the Dexcom Clarity cloud.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in normal glucose control (defined as glucose levels between 70 mg/dL - 120 mg/dL) over a seven-day period | 7 days

SECONDARY OUTCOMES:
Total number of low glycemic events (< 70 mg/dL) over a seven-day period | 7 days
Percentage of time where low glucose values were (< 70mg/dL) over a seven-day period | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (2):
- UT Health - McGovern Medical School, Houston, Texas, United States
- University Medical Center Groningen, Groningen, Netherlands